CLINICAL TRIAL: NCT02491658
Title: A Study to Assess Safety and Efficacy of Umbilical Cord Derived Mesenchymal Stem Cells (UC-MSCs) in Patients With Psoriasis Vulgaris
Brief Title: Safety and Efficacy of UC-MSCs in Patients With Psoriasis Vulgaris
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-PV-MSC
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treat Psoriasis Vulgaris with UC-MSCs (Experimental): Subjects in this arm will receive 6 times UC-MSCs infusions (each time 1×10^6/kg) within 8 weeks.
  Interventions: Biological: UC-MSCs

INTERVENTIONS:
Biological: UC-MSCs — Psoriasis Vulgaris patients will receive 6 times UC-MSCs infusions (each time 1×10^6/kg). The first time to fourth time will be given once a week for successive 4 weeks, then the last two times will be given once every two weeks.
  Other Names: umbilical cord derived mesenchymal stem cells

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of umbilical cord derived mesenchymal stem cells (UC-MSCs) in patients with moderate to severe psoriasis vulgaris. Any adverse events related to UC-MSCs infusion will be monitored and the patients will be assessed by Psoriasis Activity and Severity Index (PASI) and Dermatology Life Quality Index (DLQI) in the baseline and after MSCs infusions.

DETAILED DESCRIPTION:
Psoriasis is considered as an incurable immune-mediated inflammatory skin disease. The widely used treatments include topical agents, systemic medications and biologic agents, but all of them have some drawbacks or limitations. Besides, non-standardized treatment or the disease itself may lead transformation to other diseases, which add more importance to finding improved management strategies.

Mesenchymal stem cells (MSCs) are a heterogeneous population of cells that can differentiate into bone, cartilage and fat cells. They have several functions, such as migration to skin lesions, immunomodulation, limitation of autoimmunity and local paracrine effects. It reported MSCs have already been used in some kinds of autoimmune disease, such as systemic lupus erythematosus (SLE), systemic sclerosis, crohn disease, rheumatoid arthritis et al.

In this study, consenting umbilical cords are donated by healthy donors. After several processing steps, UC-MSCs are separated and froze for future infusions. When volunteers are recruited, their condition will be assessed by Psoriasis Activity and Severity Index (PASI) and Dermatology Life Quality Index (DLQI). Then MSCs will be infused according to a standard scheme. After all 6 infusions, the patient will be re-assessed by the PASI and DLQI and will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable psoriasis vulgaris for at least 6 months
* Baseline Psoriasis Area and Severity Index (PASI) score >= 8
* Despite systemic or topical treatment, psoriasis is still in active or recurrent condition
* No other psoriasis management (topical or systemic) during the UC-MSCs infusions
* Willing and able to comply with all study requirements and provide informed consent

Exclusion Criteria:

* Other types of psoriasis, such as pustular psoriasis, psoriatic arthritis
* With other disease
* Systemic treatments within 4 weeks before the baseline visit
* Topical treatment within 2 weeks before the baseline visit
* Uncontrolled active infections
* Evidence of infection with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV)
* History of severe systemic disease or malignancy
* Pregnant or lactating females, or willing to have a baby in the next year
* Cannot be traced on time
* Any other situations not suitable for this study determined by the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Psoriasis Area and Severity Index (PASI) score at 8 weeks | baseline and 8 weeks
  PASI score will be assessed at baseline (pre-infusion) and week 8 (right after the sixth UC-MSCs infusion)
Change from Baseline in Dermatology Life Quality Index (DLQI) score at 8 weeks | baseline and 8 weeks
  DLQI score will be assessed at baseline (pre-infusion) and week 8 (right after the sixth UC-MSCs infusion)

SECONDARY OUTCOMES:
body temperature will be monitored for any possible infusion-related toxicities. | up to 3 months
blood pressure will be monitored for any possible infusion-related toxicities. | up to 3 months
Psoriasis Area and Severity Index (PASI) score | month 6, 9, and 12
  PASI score will be assessed at month 6, 9 and 12 from the first UC-MSC infusion as followed-up.
Dermatology Life Quality Index (DLQI) score | month 6, 9, and 12
  DLQI score will be assessed at month 6, 9 and 12 from the first UC-MSC infusion as followed-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hu, Ph.D, Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China